CLINICAL TRIAL: NCT06714214
Title: PREdiction of succeSSful weanING From Continuous Renal Replacement Theraphy: the Possible Role of Delta C-cistatin
Acronym: PRESSING
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PRESSING
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-09

CONDITIONS: Acute Kidney Injury
Keywords: C cistatin; acute kidney injury; CRRT; weaning
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples With DNA — Blood to dose c-cistatin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to know if, in patients with acute kidney injury, naive for renal injurie, admitted to different ICUs, the change in plasma concentration of c-cistatin, between initiation and discontinuation of CRRT, is a predictive finding to optimize the withdrawal time of renal support

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* diagnosis of acute kidney injury (defined according to KDIGO 2012 criteria)
* need for support with CRRT according to the indications of the nephrologist consultants and Clinical Practice
* Obtaining informed consent

Exclusion Criteria:

* CRRT already ongoing (in another department not participating in the study) at the time of transfer/admission to intensive care;
* need for RRT (any type and modality) in the 14 days prior to enrolment;
* diagnosis of AKD/CKD/ESRF on admission;
* Discontinuation of CRRT under conditions that do not comply with the criteria established by the study;
* Need for CRRT not associated with AKI condition (e.g. elimination of toxicants);
* pregnant women;
* presence of known thyreopathy
* Continuous use of corticosteroids
* patient with known neoplastic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all adult patients suffering from acute renal injury needing to CRRT, admitted to the enrolling centers starting from the approval of the Ethics Committee
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
the change in plasma concentration of c-cistatin between initiation and discontinuation of CRRT is a predictive finding in patients with acute kidney injury admitted to the ICU | From enrlollment to the weaning from CRRT and 14 days after
  To verify whether the change in plasma concentration of c-cistatin between initiation and discontinuation of CRRT is a predictive finding in patients with acute kidney injury admitted to the ICU It is measured as (cistatin at weaning minus cistatin basal) divided by cistatine basal, in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Marino, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Anestesia e Terapia Intensiva nelle emergenze locali, regionali e nazionale e nella chirurgia addominale maggiore, Bologna
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna -Anestesiologia e terapia intensiva polivalente, Bologna